CLINICAL TRIAL: NCT03860610
Title: TEPStabil - Muscle Function and Dynamic and Postural Stability in Patients Receiving Hip or Knee Arthroplasty
Acronym: TEPStabil
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02159; ch19Muendermann
Record Dates: First submitted 2019-02-26; First posted 2019-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Postural Stability
Keywords: Total Hip Arthroplasty; Total Knee Arthroplasty; Osteoarthritis; Muscle strength deficits; Dynamic stability
MeSH Terms: conditions — Osteoarthritis | interventions — Range of Motion, Articular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patient group 1 after THA: Patients who have already received a THA (N=30) for OA will be assessed 1 year postoperatively (Visit A); Interventions in this Group: 'Muscle strength test', 'Dynamic stability test during level and uphill walking', 'Postural stability test', 'EuroQol Group Health questionnaire (EQ-5D-5L)', 'HOOS/ KOOS', ' Muscle activity test', 'Passive range of motion'
  Interventions: Diagnostic Test: Muscle strength test; Diagnostic Test: Dynamic stability test during level and uphill walking; Diagnostic Test: Postural stability test; Diagnostic Test: EuroQol Group Health questionnaire (EQ-5D-5L); Diagnostic Test: HOOS/ KOOS; Diagnostic Test: Muscle activity test; Diagnostic Test: Passive range of motion
- Patient group 2 after TKA: Patients who have already received a TKA (N=30) for OA will be assessed 1 year postoperatively (Visit A); Interventions in this Group: 'Muscle strength test', 'Dynamic stability test during level and uphill walking', 'Postural stability test', 'EuroQol Group Health questionnaire (EQ-5D-5L)', 'HOOS/ KOOS', ' Muscle activity test', 'Passive range of motion'
  Interventions: Diagnostic Test: Muscle strength test; Diagnostic Test: Dynamic stability test during level and uphill walking; Diagnostic Test: Postural stability test; Diagnostic Test: EuroQol Group Health questionnaire (EQ-5D-5L); Diagnostic Test: HOOS/ KOOS; Diagnostic Test: Muscle activity test; Diagnostic Test: Passive range of motion
- Patient group 3 before THA: Patients with severe hip OA (N=30) scheduled to receive a THA will be assessed preoperatively (Visit 1), 12 weeks postoperative (Visit 2) and 1 year postoperative (Visit 3). Interventions in this Group: 'Muscle strength test', 'Dynamic stability test during level and uphill walking', 'Postural stability test', 'EuroQol Group Health questionnaire (EQ-5D-5L)', 'HOOS/ KOOS', ' Muscle activity test', 'Passive range of motion'
  Interventions: Diagnostic Test: Muscle strength test; Diagnostic Test: Dynamic stability test during level and uphill walking; Diagnostic Test: Postural stability test; Diagnostic Test: EuroQol Group Health questionnaire (EQ-5D-5L); Diagnostic Test: HOOS/ KOOS; Diagnostic Test: Muscle activity test; Diagnostic Test: Passive range of motion
- Patient group 4 before TKA: Patients with severe knee OA (N=30) scheduled to receive a TKA will be assessed preoperatively (Visit 1), 12 weeks postoperative (Visit 2) and 1 year postoperative (Visit 3). Interventions in this Group: 'Muscle strength test', 'Dynamic stability test during level and uphill walking', 'Postural stability test', 'EuroQol Group Health questionnaire (EQ-5D-5L)', 'HOOS/ KOOS', ' Muscle activity test', 'Passive range of motion'
  Interventions: Diagnostic Test: Muscle strength test; Diagnostic Test: Dynamic stability test during level and uphill walking; Diagnostic Test: Postural stability test; Diagnostic Test: EuroQol Group Health questionnaire (EQ-5D-5L); Diagnostic Test: HOOS/ KOOS; Diagnostic Test: Muscle activity test; Diagnostic Test: Passive range of motion
- Healthy control group: Age-matched healthy control subjects (N=30);Interventions in this Group: 'Muscle strength test', 'Dynamic stability test during level and uphill walking', 'Postural stability test', 'EuroQol Group Health questionnaire (EQ-5D-5L)', 'HOOS/ KOOS', ' Muscle activity test', 'Passive range of motion'
  Interventions: Diagnostic Test: Muscle strength test; Diagnostic Test: Dynamic stability test during level and uphill walking; Diagnostic Test: Postural stability test; Diagnostic Test: EuroQol Group Health questionnaire (EQ-5D-5L); Diagnostic Test: HOOS/ KOOS; Diagnostic Test: Muscle activity test; Diagnostic Test: Passive range of motion

INTERVENTIONS:
Diagnostic Test: Muscle strength test — Muscle strength in knee flexion and extension and hip abduction will be tested using using a dynamometer (Biodex System 4 Pro: Biodex Medical Systems, Shirley, NY, USA)
Diagnostic Test: Dynamic stability test during level and uphill walking — Instrumented gait analysis on an overground walkway with two embedded force plates (Kistler force plate 9260AA6, Kistler AG, Winterthur, Switzerland; sampling rate 2400 Hz) and on a treadmill with an embedded plantar pressure plate (h/p/cosmos, Zebris FDM-T, Isny, Germany)
Diagnostic Test: Postural stability test — The overall stability index (OSI) will be assessed using the Biodex Balance System SD (Biodex Medical Systems, Inc., Shirley, NY, USA) and is determined by the variance in platform displacement from the horizontal plane.
Diagnostic Test: EuroQol Group Health questionnaire (EQ-5D-5L) — Overall health will be assessed using the EQ-5D-5L health questionnaire
Diagnostic Test: HOOS/ KOOS — Site specific pain and function will be assessed with the Hip Osteoarthritis Outcome Score (HOOS) and Knee Injury and Osteoarthritis Outcome Score (KOOS) depending on the affected joint (hip or knee).
Diagnostic Test: Muscle activity test — Surface electrodes (Ag/AgCl, Noraxon, U.S.A. Inc., Scottsdale, AZ, USA: 10 mm diameter, 22 mm inter-electrode distance) will be placed bilaterally on glutaeus medius, vastus medialis, semitendinosus, tibialis anterior, gastrocnemius medialis, and peroneus longus muscles. Periods of muscle activity will be defined as intensity above 2 Standard Deviation (SD) of the resting Electromyography (EMG) signal. Duration of overlapping muscle activity between agonists and antagonists normalized to one gait cycle or of a balance test, respectively, will be determined.
Diagnostic Test: Passive range of motion — Passive range of motion will be assessed for ankle plantar-/dorsiflexion, knee flexion/extension and hip flexion/extension, ab/adduction, internal/external rotation using goniometers and recorded in degrees. The range between two maxima will be recorded.

SUMMARY:
Study 1 is to determine if muscle strength and dynamic and postural stability are compromised in patients with severe hip or knee Osteoarthritis (OA) and in patients after THA and TKA.

Study 2 is to quantify the effect of THA and TKA on muscle strength and dynamic and postural stability.

DETAILED DESCRIPTION:
Postural stability is defined as the ability to maintain the body's centre of gravity within the limits of stability as determined by the base of support. It is further divided in static and dynamic stability involving the ability of maintaining a base of support while standing or completing a functional Task. The importance of postural stability is accepted as a factor predicting falls and affecting the ability to perform activities of daily living.

Despite of reported strength deficits and the importance of balance, to date the potential contribution of strength deficits in patients before and after Total Hip Arthroplasty (THA) or Total Knee Arthroplasty (TKA) to compromised balance ability is unknown. Furthermore, the role of preoperative muscle function on functional outcome of THA and TKA is poorly understood. A correlation between compromised preoperative muscular function and postoperative outcome would suggest that preoperative physical therapy may be critical for preserving the muscular status and may help explain reported poorer outcome after late treatment when muscular function has already deteriorated.

The project includes two studies differing in design and primary and secondary objectives but with overlapping patient populations.

Study 1 will include all five groups, and there is only one visit by the participant (visit A).

Study 2 will include only patients from groups 3 and 4. Three assessments will be performed: preoperatively (visit 1), 6 weeks postoperatively (visit 2) and 1 year postoperative (visit 3). Visit 1 will be identical to visit A in study 1 in these two patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an unilateral THA or TKA, which they received for the treatment of osteoarthritis (Patient groups 1+2)
* Patients diagnosed with unilateral OA of the knee or hip planned for a treatment with THA or TKA (Patient groups 3+4)
* Age ≥ 30 years (Healthy control group)

Exclusion Criteria:

* Body mass index > 35kg/m2
* Use of walking aids
* Neuromuscular disorders affecting gait
* Inability to follow procedures due to psychological disorders or dementia
* Diagnosed hip or knee OA (Healthy control group)
* Current pain in the lower extremities or lower back (Healthy control group)
* Rheumatoid Arthritis (Healthy control group)
* Previous corrective osteotomy (Healthy control group)
* Regular intake of pain medication (more than 4 times per week) (Healthy control group)

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited by consecutive recruitment through the contributing surgeons in daily clinical practice, referring physicians and advertisements placed bi-monthly in the University of Basel "Uni-news" and ongoing on the department website. Healthy participants will be recruited by advertisements placed bi-monthly in the University of Basel "Uni-news", local health and sports clubs and ongoing on the department website.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Muscle strength (Study 1) | single point measurement at Visit A (week 0)
  For the knee, maximum isokinetic flexion and extension torques will be collected between full extension and 90° flexion at a movement speed of 60°/s (5 repetitions) and 240°/s (5 repetitions).For the hip, maximum abduction torques will be measured isometrically (5 repetitions) in a standing position. Maximum joint torques in each movement direction will be recorded for each joint and normalized to body weight (study group 1 to 5)
Change in Muscle strength (Study 2) | Three assessments will be performed: preoperatively (visit 1), 6 weeks postoperatively (visit 2) and 1 year postoperative (visit 3).
  For the knee, maximum isokinetic flexion and extension torques will be collected between full extension and 90° flexion at a movement speed of 60°/s (5 repetitions) and 240°/s (5 repetitions).For the hip, maximum abduction torques will be measured isometrically (5 repetitions) in a standing position. Maximum joint torques in each movement direction will be recorded for each joint and normalized to body weight (study group 3 and 4)
Postural stability (Study 1) | single point measurement at Visit A (week 0)
  The overall stability index (OSI) will be assessed using the Biodex Balance System SD. A high stability index represents the angular excursion of the subject's center of gravity and is indicative of a high degree of movement during a test (i.e.poor balance). (study group 1 to 5)
Change in postural stability (Study 2) | Three assessments will be performed: preoperatively (visit 1), 6 weeks postoperatively (visit 2) and 1 year postoperative (visit 3).
  The overall stability index (OSI) will be assessed using the Biodex Balance System SD. A high stability index represents the angular excursion of the subject's center of gravity and is indicative of a high degree of movement during a test (i.e.poor balance).(study group 3 and 4)
Dynamic stability (Study 1) | single point measurement at Visit A (week 0)
  Instrumented gait analysis on an overground walkway to compute step width for each step from a pressure plate built into the treadmill (study group 1 to 5)
Change in dynamic stability (Study 2) | Three assessments will be performed: preoperatively (visit 1), 6 weeks postoperatively (visit 2) and 1 year postoperative (visit 3).
  Instrumented gait analysis on an overground walkway to compute step width for each step from a pressure plate built into the treadmill (study group 3 and 4)

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, Prof. Dr. MD, Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland